CLINICAL TRIAL: NCT07360418
Title: A Prospective Multicenter Study Evaluating the Durability of Closure for Diabetic Foot Ulcers Following a Randomized, Controlled, Modified Platform Trial
Brief Title: Evaluating the Durability of Closure for Diabetic Foot Ulcers Following a Randomized, Controlled, Modified Platform Trial.
Acronym: SCANX
Status: Recruiting | Type: Observational
Sponsor: Applied Biologics, LLC (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00084454
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Foot Ulcers (DFU); Foot Ulcer Chronic; Ulcer; Diabetic Foot Ulcer
Keywords: CAMPX; CAMP; Foot Ulcer; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot; Ulcer; Foot Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OneStep Foot Scanner: This study is a follow-up durability trial from the CAMPX randomized controlled clinical trial. Only subjects who achieved complete closure at 12 weeks in the CAMPX trial will be evaluated. After signing the IRB-approved informed consent form, the subject will receive instruction on the BlueDrop® OneStep Foot Scanner™. In addition, written instructions on use will be provided. Subjects that are unable to use the scale will be asked to answer a questionnaire at 3, 6, 9, and 12 months after signing the consent form.
  Interventions: Other: Blue Drop Foot Scanner

INTERVENTIONS:
Other: Blue Drop Foot Scanner — Subjects with eligible wound will receive a BlueDrop® OneStep Foot Scanner™. They are instructed to step on the scale each morning. The Bluetooth technology transmits a photograph and thermal image to the central monitoring nurse at BlueDrop®. All information transmitted is compliant with HIPPA regulations. Subjects that are unable to use the scale will receive a phone call at months 3,6, 9 and 12 months to determine if the foot has remained closed.

SUMMARY:
Prospective long-term follow-up on durability of closure evaluated by photographic and thermal scanning.

DETAILED DESCRIPTION:
This study is a follow-up durability trial from the CAMPX randomized controlled clinical trial. Only subjects who achieved complete closure at 12 weeks in the CAMPX trial will be evaluated. After signing the IRB-approved informed consent form, the subject will receive instruction on the BlueDrop® OneStep Foot Scanner™. In addition, written instructions on use will be provided. Subjects that are unable to use the scale will be asked to answer a questionnaire at 3, 6, 9, and 12 months after signing the consent form..

ELIGIBILITY:
Inclusion Criteria:

* The potential subject must have participated in the CAMPX trial and achieved complete closure by the 12-week endpoint.

Exclusion Criteria:

* The potential subject did not participate in the CAMPX trial.
* The potential subject participated in the CAMPX trial and did not achieve complete closure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from diabetic subjects who have previously completed the CAMPX trial and achieved complete closure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Recurrence | 52 weeks
  To demonstrate durability of closure (rate of recurrence) of subjects with a closed diabetic foot ulcer during the CAMPX clinical trial comparing subjects treated with Single Layer Amniotic Membrane (SLAM) plus standard of care (SOC) to subjects treated with SOC alone.

SECONDARY OUTCOMES:
Virtual Long-Term Follow Up | 52 weeks
  To evaluate the effectiveness of virtual clinical trial technology in the conduct of a long-term follow up trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Foot and Ankle, Clinton Township, Michigan, United States

IPD SHARING:
Plan to Share IPD: No